CLINICAL TRIAL: NCT05998694
Title: Post-market Clinical Monitoring of the Safety and Efficacy of the Aortic Valve Bioprothesis "ТiAra" (T-ara)
Brief Title: Post-market Clinical Monitoring of the Safety and Efficacy of the Aortic Valve Bioprothesis
Acronym: TiAra
Status: Recruiting | Type: Observational
Sponsor: Closed Joint-Stock Company NeoCor (Other)
Collaborators: CT Medical Limited Liability Company (Unknown); Research Institute for Complex Problems of Cardiovascular Diseases, Russia (Other)
Responsible Party: Sponsor
Other Study IDs: (T-ara) TA0120
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Aortic Valve Disease; Artificial Heart Valves
Keywords: aortic valve; aortic valve bioprothesis TiAra; valve bioprosthesis; hemolysis; hemolytic anemia; a heart stroke; myocardial infarction; hemorrhaging and bleeding; heart arrhythmia; nonstructural dysfunction; pannus; prosthesis-patient mismatch; dislocation; paraprosthetic and transprosthetic regurgitation; heart failure; breast-pang; structural deterioration; valve thrombosis; thromboembolism; encarditis; a reoperation
MeSH Terms: conditions — Aortic Valve Disease; Hemolysis; Anemia, Hemolytic; Myocardial Infarction; Hemorrhage; Arrhythmias, Cardiac; Joint Dislocations; Heart Failure; Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this multicenter prospective cohort study is to evaluate the long-term safety and efficacy of clinical outcomes of aortic valve replacement using the "TiAra" prosthesis with or without concomitant procedures.

Main research objectives:

1. To analyze the short and mid-term (up to 3 years) outcome of aortic valve replacement using the "TiAra" prosthesis.
2. To study the hemodynamic characteristics of normally functioning "TiAra" prostheses in the aortic position, as well as the condition of the heart chambers in short and long-term period (up to 10 years) after the implantation.
3. To assess complications of the early and mid-term follow-up periods of aortic valve replacement using the "TiAra" prosthesis.

This study does not presuppose implementation of comparison groups.

DETAILED DESCRIPTION:
Cardiovascular system diseases are one of the main causes of death worldwide. Heart valve diseases are considered one of the most important issues associated with the cardiovascular system. The replacement of heart valves includes the production of prostheses that provide functional consistency with exceptionally high reliability and appropriate fatigue strength. The proposed new biological valve with a frame made of super-elastic material allows preserves the natural biomechanics of the reconstructed valve and has high biocompatibility and resistance to infection due to the use of biological material as a frame covering. The "TiAra" bioprosthetic valve has the ability to deform during the cardiac cycle in accordance with the deformations of the fibrous structures of the patients' aortic root. The implanted valve fully integrates into the native aortic root.

The purpose of these clinical trials is to obtain clinical data confirming the efficacy and safety of the bioprosthesis under normal conditions in humans.

The expected clinical benefit involves the treatment of valvular disease with restoration of intracardiac hemodynamics during implantation of the "TiAra" bioprosthetic valve, followed by remodeling of the heart chambers, which should lead to an improvement in heart function and quality of life of the patient.

The expected risks are associated with taking anticoagulant therapy during the first three months after implantation, or as a result of prolonged anticoagulant therapy, in the presence of concomitant rhythm disturbances, and consist in the possibility of hemorrhagic or thromboembolic complications. In order to reduce the risks caused by anticoagulant therapy, it is planned to carry out measures aimed at restoring the sinus rhythm and ensuring proper control of the indicators of the blood coagulation system.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's written consent to participate in the study and the absence of restrictions on physical movement (diseases of the musculoskeletal system and diseases of the central nervous system, accompanied by cognitive disorders (disorientation, inability to independently reach the destination).
2. The patient is a resident of the city* (suburb) where the institution is conducting study.

   * - participation is also possible for those living in the rural areas, but they have to be able to make visits to the Research Center.
3. Age: 60-70 years old with a life expectancy of 3 years or more. Or a person younger than 60 with contraindications to taking anticoagulants, or with increased risk of their use, consciously choosing a biological prosthesis for valve replacement.
4. Isolated aortic valve disease.
5. Real intervention on the heart valve is primary.
6. Absence of concomitant interventions on the heart and thoracic aorta**.

   ** - Coronary artery bypass grafting, correction of tricuspid valve disease, previously treated congenital heart defects, aortic intervention
7. The intervention on the valve is planned (that is, it is not carried out in expedited/urgent manner or is not a "rescue" operation).
8. Absence of acute and subacute infective endocarditis.
9. The following factors should not be present before surgery: high pulmonary hypertension (pulmonary arterial systolic pressure more than 60 mmHg), functional class 4 (according to the New York Heart Association Functional Classification) while in ongoing treatment, left ventricular ejection fraction less than 30%.

Exclusion Criteria:

1. The presence of severe somatic, neurological, mental diseases and infectious diseases that worsen the prognosis of long-term survival (ischemic heart disease, tuberculosis, human immunodeficiency viruses, Alzheimer's disease, epilepsy, insulin-requiring diabetes, kidney disease with creatinine clearance less than 85 mL/min, chronic lung disease requiring chronic corticosteroids and bronchodilators, multifocal atherosclerosis (intermittent claudication, carotid arteries stenosis of more than 50%, prior and planned interventions on abdominal area, carotid arteries or arteries of the lower extremities).
2. The patient has any not related to the underlying cardiovascular system disease pathology that will lead to the death of the patient in less than 1 year.
3. The patient is currently participating in a study of a new drug or other medical devices.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As part of these clinical trials (studies), the use of comparison groups is not planned.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
1. Incidence of Treatment-Emergent Adverse Events, requiring repeated surgical intervention in the long term (long-term safety and durability) | Up to 12 years from the moment of implantation .
  Long-term safety of the "TiAra" epoxy-treated prosthesis made with xenopericardium will be evaluated by the frequency of complications associated with the valve.
  Device safety is defined as the absence of severe adverse events associated with the device or procedure, assessed by the following clinical phenomena:
  Death Severe complications of the heart Life-threatening bleeding Any bioprosthesis-related dysfunction, migration, thrombosis or other complication requiring an open-heart surgery or repeated intervention.
  Myocardial infarction or progression of a chronic form of ischemia requiring percutaneous coronary intervention and coronary artery bypass grafting Access site complications Stroke
2. Incidence of Treatment-Emergent Adverse Events, requiring repeated surgical intervention in the short term (short-term safety) | Up to 12 years from the moment of implantation
  Short-term safety of the "TiAra" epoxy-treated prosthesis made with xenopericardium in the treatment of isolated mitral and aortic valve diseases will be evaluated by the frequency of complications associated with the valve.
  Device safety is defined as the absence of severe adverse events associated with the device or procedure, assessed by the following clinical phenomena:
  hemolysis hemolytic anemia a heart stroke myocardial infarction hemorrhaging and bleeding heart arrhythmia nonstructural dysfunction pannus prosthesis-patient mismatch dislocation paraprosthetic and transprosthetic regurgitation heart failure breast-pang structural deterioration valve thrombosis thromboembolism encarditis a reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Evtushenko, MD,PhD, Principal Investigator — Research Institute for Complex Problems of Cardiovascular Diseases, Russia
Locations (1):
- Research Institute for Complex Problems of Cardiovascular Diseases, Russia, Kemerovo, Kemerovo Oblast, Russia